CLINICAL TRIAL: NCT00809575
Title: Prognostic Significance and Longitudinal Assessment of Patient-reported Quality of Life and Symptoms in Myelodysplastic Syndromes. A Large-scale International, Observational Study: PROMYS Study
Brief Title: Quality of Life and Symptoms in Patients With Newly Diagnosed Myelodysplastic Syndromes
Acronym: PROMYS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: QOL-MDS0108; GIMEMA-QOL-MDS-0108; EU-20885; NCT00872768 (obsolete NCT alias)
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Adult; Myelodysplastic Syndromes
Keywords: adult; de novo myelodysplastic syndromes; Quality of life; Patient reported outcomes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Therapeutics; Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: questionnaire administration
Other: fatigue assessment and management
Other: observation
Other: quality-of-life assessment

SUMMARY:
RATIONALE: Gathering information about quality of life, fatigue, and other symptoms from patients with myelodysplastic syndromes may help doctors learn more about the disease and may help plan treatment.

PURPOSE: This clinical trial is studying quality of life and symptoms in patients with newly diagnosed myelodysplastic syndromes.

DETAILED DESCRIPTION:
This study will ultimately aim at providing the scientific community with additional patient-reported health status data to support and further facilitate the clinical decision-making process. This project has thus a number of goals. The main objective of the protocol is to improve our understanding of the possible added prognostic value of patients' judgment on their own health status and its potential clinical implications. This would aim at providing clinicians with an easy and brief to administer patient-reported health status scale or tool to be used to make more informed treatment decisions. In addition, along with other recent evidence (also looking at the prognostic value of patients' health status judgment in MDS patients), the data of this research could possibly serve to devise a patient-based prognostic index to be used in this higher risk population.

ELIGIBILITY:
Inclusion criteria

* Patients with newly diagnosed myelodysplastic syndrome (MDS) according to WHO classification with any known IPSS risk score category. The initial diagnosis of MDS is acceptable within 3 months before date of registration.
* Having a full baseline QoL Evaluation completed (i.e. EORTC QLQ-C30; EQ5D; FACIT-Fatigue and Control Preference Scale).
* Adult patients (≥ 18 years old).
* Written informed consent provided.

Exclusion criteria

* Patients who have received prior treatment other than platelets or RBC transfusions, iron chelation, antibiotic/virostatic drugs, vitamins;
* Patients with therapy related MDS.
* Having any kind of psychiatric disorder or major cognitive dysfunction.
* Not able to read and understand local language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with myelodysplastic syndromes (MDS).
Sampling Method: Non-Probability Sample
Enrollment: 927 (Actual)
Dates: Start 2008-10-02 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
To investigate the prognostic value of baseline patients' reported fatigue for overall survival in newly diagnosed myelodysplastic syndrome (MDS) patients. | After 5 years from study entry.

SECONDARY OUTCOMES:
To investigate the prognostic value of changes overtime of QoL and symptoms for clinical outcomes. | After 5 years from study entry.
  i.e. overall survival, AML transformation, toxicity and response to therapy.
To describe prospectively short and long-term symptom burden and QoL outcomes by risk group and by type of therapy. | After 5 years from study entry.
To compare the QoL of lower risk patients who maintain stable disease versus those who have progressed to AML or higher-risk score categories. | After 5 years from study entry.
To compare the QoL and symptoms baseline reference data to be used as benchmarks for comparisons in clinical trials. | After 5 years from study entry.
To establish international QoL and symptoms baseline reference data to be used as benchmarks for comparisons in clinical trials. | After 5 years from study entry.
To evaluate the impact of transfusion dependency at baseline and over time on survival and QoL outcomes. | After 5 years from study entry.
To devise a prognostic patient-based index. | After 5 years from study entry.
To evaluate accuracy of clinical prediction of survival. | After 5 years from study entry.
To assess patients' preferences for involvement in treatment decision-making across different risk group and examine relationships between preferences and patient characteristics. | After 5 years from study entry.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Efficace, PhD, Principal Investigator — Gruppo Italiano Malattie EMatologiche dell'Adulto
Locations (53):
- United States (2):
  - Memorial Sloan-Kettering Cancer Center (MSKCC), New York, New York
  - The University of Texas, MD Anderson Cancer Center, Houston, Texas
- Innsbruck University Hospital, Innsbruck, Austria
- Belgium (4):
  - ZNA Middelheim, Antwerp
  - AZ Sint-Jan AV, Department of Hematology, Bruges
  - CH Jolimont, Brussels
  - CHC - Centre Hospitalier Chrétien, Liège
- Curitiba Unidade de Hematologia - Hemoterapia e Oncologia. Setor de Transplante de Medula Ossea. Complexo Hospital de Clinicas da Universidade Federal do Parana (CHC-UFPR), Curitiba, Brazil
- China (2):
  - Affiliated Hospital of Liaoning University of Traditional Chinese Medicine, China
  - Kunming Medical University, Kunming
- Hematology - Clinical Hospital Centre Rijeka - Faculty of Medicine - University of Rijeka, Rijeka, Croatia
- General Teaching Hospital, Prague, Czechia
- France (2):
  - Saint - Cloud Medecin des CLCC Hematologie Service E Hopital ReneHuguenin - Institut Curie, Saint-Cloud
  - Purpan Hospital - Internal Medicine Department, Toulouse
- Germany (2):
  - Department of Hematology - Universitatsklinikum Carl Gustav Carus, Dresden
  - University of Freiburg Medical Center, Freiburg im Breisgau
- Italy (33):
  - Istituto di Ematologia - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - U.O.A. di Medicina Trasfusionale e DH di Ematologia - ASL TO 4 Ospedale di Ivrea, Ivrea, Torino
  - Asl Di Asti - Ospedali Riuniti - Presidio Ospedaliero Cardinal G. Massaia - Sc Oncologia, Asti
  - Unità Operativa Ematologia 1 - Università degli Studi di Bari, Bari
  - ASL N.8 - Ospedale "A. Businco" - Unità Operativa di Ematologia e Trapianto di Midollo, Cagliari
  - CTMO - Ematologia - Ospedale "Binaghi", Cagliari
  - Ospedale "Ferrarotto", Catania
  - A.O. Pugliese Ciaccio, Catanzaro
  - Aou Arcispedale Sant'Anna - Uoc Ematologia E Fisiopatologia Della Coagulazione, Cona
  - Aou Careggi - Firenze - Sod Ematologia, Florence
  - Divisione Ematologia - Azienda Ospedaliera Universitaria "San Martino"", Genova
  - Divisione di Ematologia Ospedale "Santa Maria Goretti", Latina
  - ASL Le1 P.O. Vito Fazzi - U.O. di Ematologia, Lecce
  - Istituto Scientifico Romagnoli per lo Studio e la Cura dei Tumori- IRST, Meldola
  - U.O. Ematologia e Trapianto di Midollo - Ist. Scientifico Ospedale San Raffaele, Milan
  - Ospedale Niguarda "Ca Granda", Milan
  - UO Ematologia - AOU Policlinico di Modena, Modena
  - Asst Di Monza - Ospedale S. Eugenio - Uo Ematologia E Cta, Monza
  - S.C.D.U. Ematologia - DIMECS e Dipartimento Oncologico - Università del Piemonte Orientale Amedeo Avogadro, Novara
  - Ospedale S. Luigi Gonzaga, Orbassano
  - Aou Di Parma - Sc Ematologia E Centro Trapianti Midollo Osseo, Parma
  - Med. Int. ed Oncologia Medica IRCCS Policlinico S. Matteo, Pavia
  - Asl Di Piacenza - Ospedale "Guglielmo Da Saliceto" - Ematologia E Centro Trapianti, Piacenza
  - Ausl Di Reggio Emilia - Arcispedale Santa Maria Nuova - Irccs - Sc Ematologia, Reggio Emilia
  - Divisione Ematologia - Università Campus Bio-Medico, Roma
  - Università degli Studi - Policlinico di Tor Vergata, Roma
  - Università degli Studi "La Sapienza" - Dip. Biotecnologie Cellulari ed Ematologia - Divisione di Ematologia, Roma
  - Università Cattolica del Sacro Cuore - Policlinico A. Gemelli, Roma
  - Complesso Ospedaliero S. Giovanni Addolorata, Roma
  - U.O.C. Ematologia - Ospedale S.Eugenio, Rome
  - SOS Dipartimento di Oncoematologia Osp. Rovigo, Rovigo
  - Ematologia - Dipartimento di Medicina Clinica e Sperimentale, Sassari
  - Aou Città Della Salute E Della Scienza - Ospedale S. Giovanni Battista Molinette, Torino
- National Taiwan University, Taipei, Taiwan
- United Kingdom (3):
  - Bradford Institute of Health Research, Bradford
  - St James's University Hospital, Leeds
  - London North West Healthcare NHS Trust, London

REFERENCES:
- [Background] Efficace F, Gaidano G, Sprangers M, Cottone F, Breccia M, Voso MT, Caocci G, Stauder R, Di Tucci AA, Sanpaolo G, Selleslag D, Angelucci E, Platzbecker U, Mandelli F. Preference for involvement in treatment decisions and request for prognostic information in newly diagnosed patients with higher-risk myelodysplastic syndromes. Ann Oncol. 2014 Feb;25(2):447-54. doi: 10.1093/annonc/mdt557. PMID 24478321
- [Background] Caocci G, Voso MT, Angelucci E, Stauder R, Cottone F, Abel G, Nguyen K, Platzbecker U, Beyne-Rauzy O, Gaidano G, Invernizzi R, Molica S, Criscuolo M, Breccia M, Lubbert M, Sanpaolo G, Buccisano F, Ricco A, Palumbo GA, Niscola P, Zhang H, Fenu S, La Nasa G, Mandelli F, Efficace F. Accuracy of physician assessment of treatment preferences and health status in elderly patients with higher-risk myelodysplastic syndromes. Leuk Res. 2015 Aug;39(8):859-65. doi: 10.1016/j.leukres.2015.05.012. Epub 2015 Jun 12. PMID 26120100
- [Background] Efficace F, Gaidano G, Breccia M, Criscuolo M, Cottone F, Caocci G, Bowen D, Lubbert M, Angelucci E, Stauder R, Selleslag D, Platzbecker U, Sanpaolo G, Jonasova A, Buccisano F, Specchia G, Palumbo GA, Niscola P, Wan C, Zhang H, Fenu S, Klimek V, Beyne-Rauzy O, Nguyen K, Mandelli F. Prevalence, severity and correlates of fatigue in newly diagnosed patients with myelodysplastic syndromes. Br J Haematol. 2015 Feb;168(3):361-70. doi: 10.1111/bjh.13138. Epub 2014 Oct 1. PMID 25272332
- [Background] Efficace F, Gaidano G, Breccia M, Voso MT, Cottone F, Angelucci E, Caocci G, Stauder R, Selleslag D, Sprangers M, Platzbecker U, Ricco A, Sanpaolo G, Beyne-Rauzy O, Buccisano F, Palumbo GA, Bowen D, Nguyen K, Niscola P, Vignetti M, Mandelli F. Prognostic value of self-reported fatigue on overall survival in patients with myelodysplastic syndromes: a multicentre, prospective, observational, cohort study. Lancet Oncol. 2015 Nov;16(15):1506-1514. doi: 10.1016/S1470-2045(15)00206-5. Epub 2015 Sep 21. PMID 26404501
- [Background] Efficace F, Cottone F, Abel G, Niscola P, Gaidano G, Bonnetain F, Anota A, Caocci G, Cronin A, Fianchi L, Breccia M, Stauder R, Platzbecker U, Palumbo GA, Luppi M, Invernizzi R, Bergamaschi M, Borin L, Di Tucci AA, Zhang H, Sprangers M, Vignetti M, Mandelli F. Patient-reported outcomes enhance the survival prediction of traditional disease risk classifications: An international study in patients with myelodysplastic syndromes. Cancer. 2018 Mar 15;124(6):1251-1259. doi: 10.1002/cncr.31193. Epub 2017 Dec 12. PMID 29231969
- [Background] Efficace F, Cottone F, Oswald LB, Cella D, Patriarca A, Niscola P, Breccia M, Platzbecker U, Palumbo GA, Caocci G, Stauder R, Ricco A, Petranovic D, Caers J, Luppi M, Fianchi L, Frairia C, Capodanno I, Follini E, Sarlo C, Fazi P, Vignetti M. The IPSS-R more accurately captures fatigue severity of newly diagnosed patients with myelodysplastic syndromes compared with the IPSS index. Leukemia. 2020 Sep;34(9):2451-2459. doi: 10.1038/s41375-020-0746-8. Epub 2020 Feb 21. PMID 32086447